CLINICAL TRIAL: NCT06966063
Title: Additive Effects of 4-7-8 Breathing Technique With Standard Management on Dyspnea, Pulmonary Function and Quality of Life in Patients With COPD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/69
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Dyspnea
Keywords: Dyspnea; pulmonary function; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Patients in interventional group will recieve 4-7-8 breathing along with standard management.
  For 4-7-8 breathing, Patient is asked sit in comfortable position. Patient is asked place the tip of your tongue up against the back of your front teeth. Keep it there through the entire breathing process. Instruct the patient to breathe in silently through your nose to the count of four (4sec) and Hold your breath to the count of seven (7sec). Exhale through your mouth to the count of eight (8sec), making an audible "whoosh" sound. That completes one full breath. Repeat the cycle another three time, and gradually in increase the cycle four time.
  Total 4 weeks protocol. Two sessions per week will be supervised by physiotherapist and 5 days at home. A home diary will be provided in order to ensure and follow-up that participants are performing breathing exercise at home along with medications prescribed by pulmonologist.
  Interventions: Procedure: 4-7-8 breathing along with standard management.
- Control group (Active Comparator): Patients will receive medication as prescribed by pulmonologist through stepwise approach according to symptoms and severity.
  Total 4 weeks protocol. Before and after 4 weeks pre and post interventional values will be taken.
  Week 01 and 02 Patients will receive medications prescribed by pulmonologist. Week 03 and 04 Patients will receive medications prescribed by pulmonologist.
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: 4-7-8 breathing along with standard management. — For 4-7-8 breathing, Patient is asked sit in comfortable position. Patient is asked place the tip of your tongue up against the back of your front teeth. Keep it there through the entire breathing process. Instruct the patient to breathe in silently through your nose to the count of four (4sec) and Hold your breath to the count of seven (7sec). Exhale through your mouth to the count of eight (8sec), making an audible "whoosh" sound. That completes one full breath. Repeat the cycle another three time, and gradually in increase the cycle four time.
  Total 4 weeks protocol. Two sessions per week will be supervised by physiotherapist and 5 days at home. Week 01 and 02 Frequenc: 01 session/day Intensity: Start with comfortable duration. Time: 10 minutes Week 03 and 04 Frequecy: 02 sessions/day Intensity: 4 sec inhale, 7 sec hold and 8 sec exhale Time: 15 minutes
  Arms: Interventional group
Procedure: Control Group — Patients will recieve medication as prescribed by pulmonologist through stepwise approach according to symptoms and severity.
  Total 4 weeks protocol. Before and after 4 weeks pre and post interventional values will be taken.
  Week 01 and 02 Patients will receive medications prescribed by pulmonologist. Week 03 and 04 Patients will receive medications prescribed by pulmonologist.
  Arms: Control group

SUMMARY:
A heterogeneous lung condition characterized by chronic respiratory symptoms (dyspnea, cough, expectoration and/or exacerbations) due to abnormalities of the airways (bronchitis, bronchiolitis) and/or alveoli (emphysema)-- cause persistent, often progressive, airflow obstruction.

Breathing exercises help to manage dyspnea and reduced pulmonary function often seen in COPD patients. To handle respiratory complications COPD patients are advised to practice breathing techniques in conjunction with their prescribed medications.

DETAILED DESCRIPTION:
COPD is a very common chronic respiratory disease with symptoms (dyspnea, cough, expectoration and/or exacerbations) due to abnormalities of the airways (bronchitis, bronchiolitis) and/or alveoli (emphysema)-- cause persistent, often progressive, airflow obstruction.

Breathing exercises help to manage dyspnea associated with COPD. In order to manage respiratory conditions COPD patients are encouraged for nasal breathing techniques along with standard management. Hence the objective of the study is to compare the effects of 4-7-8 breathing along with standard management versus standard management alone on dyspnea, pulmonary function, and quality of life in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Adults: aged (40-64 years)
* Gender: Both males and females
* Grade1- Grade 1-3 on Modified MRC dyspnea scale
* COPD mild and moderate according to GOLD classification
* Mild: FEV1 > 80% predicted
* Moderate: FEV1 >50% predicted

Exclusion Criteria:

* Severe and very severe stage of COPD according to GOLD classification.
* Patients having Acute exacerbation of COPD.
* Patients diagnosed with acute infections.
* Patients unable to follow commands/ instructions.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Dyspnea | 4 weeks
  Evaluation will be done using Dyspnea-12 questionnaire for dyspnea
pulmonary function | 4 weeks
  spirometer to measure volume of air inspired and exhale through lungs.
Quality of Life of COPD patients | 4 weeks
  COPD assessment test (CAT) will be used to evaluate quality of life of COPD patients

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan